CLINICAL TRIAL: NCT00267397
Title: Prevalence and Clincial Spectrum of the 22q11 Deletion: A Population Based Study of Children and Congenital Heart Defects
Brief Title: Prevalence and Clinical Spectrum of the 22q11 Deletion
Status: Terminated | Type: Observational
Why Stopped: sufficient data collected
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 01-107
Record Dates: First submitted 2005-12-19; First posted 2005-12-21 (Estimated); Last update posted 2007-05-04 (Estimated); Status verified 2007-05

CONDITIONS: Congenital Disorders
Keywords: infant; prenatal; birth defects; 22Q11 deletion
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Congenital Abnormalities; DiGeorge Syndrome

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this project is to conduct population based surveillance for prenatally diagnosed congenital defects amount residents of the five counties to: improve the comprehensiveness of the Metropolitan Atlanta Congenital Defects Program (MACDP) to (1) better fulfill its objectives (2) allow assessment of the impact of prenatal diagnosis and elective termination on the birth prevalence of congenital defects in Atlanta (3) develop a registry of prenatally diagnosed defects to be used in epidemiologic and genetic studies, in evaluation prevention programs and in monitoring prenatal diagnostic technology.

DETAILED DESCRIPTION:
Since 1967, The Centers for Disease Control and Prevention (CDC) has conducted surveillance of birth defects in metropolitan Atlanta through review of hospital delivery and newborn medical records and records from various other medical sources in the five central counties of the metropolitan area (Clayton, Cobb, DeKalk, Fulton and Gwinnett, and has been expanded to include prenatal records. The project was begun n the aftermath of thalidomide and rubella epidemics as a kind of early-warning system for new or resurgent teratogens. The voluntary participation of Atlanta hospitals was sought and obtained at the inception of the system (the original system was a joint effort of the CDC, the Georgia Institute of Mental Health and Emory University).

A case must be diagnosed by the child's sixth birthday or within six years of the date of elective termination.

Children's Healthcare is one retrospective source of medical records reviewed for discharge summaries and disease indices.

ELIGIBILITY:
Inclusion Criteria:

* birth defect diagnosed by the child's sixth birthday
* birth defect diagnosed within 6 years of the elective date of termination

Exclusion Criteria:

* those who do not meet inclusion criteria

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1967-01; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Campbell, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States